CLINICAL TRIAL: NCT04236453
Title: A Single-Dose, Open-Label, Randomized, Replicate Crossover Pivotal Bioequivalence Study in Healthy Subjects to Assess the Bioequivalence of Darunavir 675 mg, Emtricitabine 200 mg, and Tenofovir Alafenamide 10 mg in the Presence of Cobicistat 150 mg When Administered as a Fixed Dose Combination (Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide) Compared to the Co-administration of the Separate Agents (Darunavir, Cobicistat, and Emtricitabine/Tenofovir Alafenamide), Under Fed Conditions
Brief Title: A Study in Healthy Participants to Assess the Effect of Darunavir, Emtricitabine, and Tenofovir Alafenamide in the Presence of Cobicistat When Administered as a Fixed Dose Combination (Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide) Compared to the Co-administration of the Separate Agents
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: COVID-19 pandemic impacted the BE assessment of the trial. The clinical team decided to terminate the trial in order to start a new pivotal BE trial
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108649; 2019-002245-37 (EudraCT Number); TMC114FD2HTX1005 (Other: Janssen Pharmaceutica N.V., Belgium)
Record Dates: First submitted 2020-01-21; First posted 2020-01-22 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Healthy
MeSH Terms: interventions — Darunavir; emtricitabine tenofovir alafenamide; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Participants will receive Treatment A (a single dose of Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide [D/C/F/TAF] as one fixed dose combination [FDC] tablet under fed condition on Day 1) as per assigned treatment sequence (Treatment sequence ABBA or BAAB). A wash out period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide FDC; Drug: Darunavir; Drug: Emtricitabine/Tenofovir Alafenamide; Drug: Cobicistat
- Treatment B (Active Comparator): Participants will receive Treatment B (a single dose of Darunavir [DRV], Emtricitabine/Tenofovir Alafenamide [F/TAF] and Cobicistat [COB] tablet under fed condition on Day 1) as per assigned treatment sequence (Treatment sequence ABBA or BAAB). A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide FDC; Drug: Darunavir; Drug: Emtricitabine/Tenofovir Alafenamide; Drug: Cobicistat

INTERVENTIONS:
Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide FDC — Participants will receive a single dose of Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide FDC tablet orally on Day 1 of treatment periods with Treatment A.
  Other Names: TMC114/JNJ-48763364/JNJ-35807551/JNJ-63625328
Drug: Darunavir — Participants will receive a single dose of Darunavir orally on Day 1 of treatment periods with Treatment B.
Drug: Emtricitabine/Tenofovir Alafenamide — Participants will receive a single dose of Emtricitabine/Tenofovir Alafenamide tablet orally on Day 1.
Drug: Cobicistat — Participant will receive a single dose of Cobicistat tablet orally on Day 1.

SUMMARY:
The purpose of the study is to evaluate the single-dose pharmacokinetics (PK) and pivotal bioequivalence of 3 compounds Darunavir (DRV), emtricitabine (FTC), and tenofovir alafenamide (TAF) in the presence of cobicistat (COBI) when administered as an fixed dose combination (FDC) (Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide [D/C/F/TAF]) compared to the co-administration as the separate commercial formulations (DRV and F/TAF and COBI), under fed conditions, in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy on the basis of physical examination, medical history, vital signs, and electrocardiogram (ECG) performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Participant must be healthy on the basis of clinical laboratory test performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant.
* A woman (of childbearing potential) must have a negative highly sensitive serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test, 4 days or less before dosing of the first treatment period
* Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for participant participating in clinical studies
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 90 days after receiving the last dose of study drug
* During the study and for a minimum of at least 90 days after receiving the last dose of study drug, a male participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person (male subject should also be advised of the benefit for a female partner to use a highly effective method of contraception as condom may break or leak); must agree not to donate sperm for the purpose of reproduction.
* Must be willing and able to adhere to the prohibitions and restrictions specified in the study protocol

Exclusion Criteria:

* Has history or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease (including bronchospastic respiratory disease), diabetes mellitus, hepatic or renal insufficiency (for example, estimated creatinine clearance below less than [<] 90 milliliter per minute [mL/min] at screening), gastrointestinal disease (such as significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability), thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Had one or more of the laboratory abnormalities at screening as outlined in the protocol by the Division of Acquired immunodeficiency syndrome (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events and in accordance with the normal ranges of the clinical laboratory
* Clinically significant abnormalities during physical examination, vital signs, or 12 lead electrocardiogram (ECG) at screening or at admission to the study center as deemed appropriate by the investigator
* With any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria
* Has a history of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-V) criteria within 1 year before screening or positive test result(s) for alcohol and/or drugs of abuse (such as hallucinogens, barbiturates, opiates, opioids, cocaine, cannabinoids, amphetamines, methadone, benzodiazepines, methamphetamine, tetrahydrocannabinol, phencyclidine, and tricyclic antidepressants) either at screening or on Day 1 of each treatment period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Analyte Concentration (Cmax) of Darunavir, Cobicistat, Emtricitabine and Tenofovir Alafenamide | Up to 72 hours post-dose
  Cmax is the maximum observed analyte concentration.
Area Under the Analyte Concentration-time Curve from time Zero to Last Quantifiable time (AUC[0-last]) of Darunavir, Cobicistat, Emtricitabine and Tenofovir Alafenamide | Up to 72 hours post-dose
  AUC(0-last) is the area under the analyte concentration-time curve of from time 0 to the time of the last measurable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.

SECONDARY OUTCOMES:
Area Under the Analyte Concentration-time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Darunavir, Cobicistat, Emtricitabine and Tenofovir Alafenamide | Up to 72 hours post-dose
  AUC (0-infinity) is the area under the analyte concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(last)/lambda(z); wherein AUC(0-last) is area under the analyte concentration-time curve from time zero to last quantifiable time, C(last) is the last observed measurable concentration, and lambda(z) is elimination rate constant.
Cmax of Cobicistat | Up to 72 hours post-dose
  Cmax is the maximum observed analyte concentration of Cobicistat.
AUC(0-last) of Cobicistat | Up to 72 hours post-dose
  AUC(0-last) is the area under the analyte concentration-time curve of from time 0 to the time of the last measurable (non-BQL) concentration, calculated by linear-linear trapezoidal summation.
Number of Participants with Adverse Events | From signing of the Informed consent form (ICF) till the last study-related activity (up to 10 weeks)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trials, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (1):
- PRA Health Sciences Onderzoekscentrum Groningen, locatie Martini, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency